CLINICAL TRIAL: NCT07008365
Title: The Role of intraABDOminal Pressure and Point Of Care UltraSound to Guide Decongestive Therapy in Heart Failure
Acronym: ABDOPOCUS-HF
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Instituto de Investigación Sanitaria Aragón (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PI23/00797
Record Dates: First submitted 2024-08-08; First posted 2025-06-06 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2024-08

CONDITIONS: Acute Heart Failure; Congestive Heart Failure; Intraabdominal Hypertension; Cardio-Renal Syndrome
Keywords: Point of care Ultrasound (POCUS); Acute Heart Failure; Cardio-renal syndrome; Intraabdominal pressure; Diuretic treatment
MeSH Terms: conditions — Heart Failure; Intra-Abdominal Hypertension; Cardio-Renal Syndrome

STUDY DESIGN:
Intervention Model Description: After conducting an initial comprehensive evaluation and confirming the inclusion and exclusion criteria, along with obtaining the necessary informed consent (screening), the patient will be randomized within the first 24 hours of admission into one of the two treatment groups with the aim of determining whether a diuretic treatment strategy based on intra-abdominal pressure and clinical ultrasound is superior to the conventional diuretic treatment strategy for resolving systemic congestion after the first 72 hours of admission.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standart of care treatment arm. (No Intervention): Loop diuretics (furosemide) will be administered intravenously according to stantard of care (Latest European heart failure guidelines)
- Treatment guided by intra-abdominal pressure values (Experimental): Decongestive treatment will be adjusted according to intraabdominal pressure values (IAP) and/or point of care ultrasound:
  Patients with IAP < 8 mmHg (normal): The intravenous diuretic dose will be twice the patient's previous oral dose. If no diuretics were taken previously, 20 mg of furosemide will be administered every 12 hours.
  Patients with IAP between 8 and 12 mmHg (moderately elevated): furosemide will be administered in combination with hydrochlorothiazide Patients wiht IAP > 12: Furosemide will be initiated as a continuous infusion along with hydrochlorothiazide
  Interventions: Drug: Furosemide 20 Milligrams

INTERVENTIONS:
Drug: Furosemide 20 Milligrams — Decongestive therapy with e.v. furosemide +/- hydrochlorothiazide will be adjusted by intraabdominal pressure and/or point of care ultrasound
  Other Names: furosemide 500 milligrams; hydrochlorothiazide 25 milligrams
  Arms: Treatment guided by intra-abdominal pressure values

SUMMARY:
Systemic venous congestion is the primary therapeutic target of intravenous loop diuretics in patients admitted for acute heart failure (AHF). Despite their utility, a significant proportion of AHF patients are discharged with persistent clinical symptoms of congestion (residual congestion). Therefore, in recent years, there has been a growing focus on the use of tools (biomarkers, clinical ultrasound) that allow us to optimize diuretic treatment and thereby improve the prognosis of AHF patients. The objective is to analyze whether the strategy of guiding intravenous loop diuretic dosing based on intra-abdominal pressure(IAP) measurements and clinical ultrasound is superior to the conventional strategy employed in daily clinical practice. This study is a randomized, multicenter clinical trial involving consecutive patients admitted with a diagnosis of AHF in the Internal Medicine and Cardiology departments. Patients who meet the inclusion criteria, after signing informed consent, will be randomized into two groups: 1) Diuretic treatment guided by usual clinical practice and 2) Treatment guided by intra-abdominal pressure levels and clinical ultrasound (inferior vena cava and portal Doppler). This strategy will be maintained during the first 72 hours of admission, with a thorough analysis of congestion and diuretic response being conducted.

ELIGIBILITY:
Inclusion Criteria:

* Men or women over 18 years of age.
* Diagnosis of heart failure (HF) based on the latest HF guidelines published in 2022.
* N-terminal pro b-type natriuretic peptide (NT-proBNP) > 1000 pg/mL or Brain Natriuretic Peptide (BNP) > 250 pg/mL.
* Placement of a urinary catheter to allow for the measurement of intra-abdominal pressure.
* Intravascular or mixed congestion pattern, defined as the presence of one or more clinical signs of congestion (edema, ascites, and/or pleural effusion).
* Signed informed consent

Exclusion Criteria:

* Patient with a stay in the Internal Medicine department > 24 hours.
* Absence of sufficient clinical congestion (ADVOR score = 0 at the time of randomization).
* Patient's refusal to participate in the clinical trial.
* Inability or contraindication for urinary catheter placement.
* Systolic blood pressure at admission < 100 mmHg.
* Heart rate at admission > 170 beats per minute (bpm).
* Cardiogenic shock.
* Acute myocardial ischemia.
* Patients receiving renal replacement therapy (ultrafiltration or peritoneal dialysis).
* Kidney transplant recipients.
* Serum hemoglobin < 9 g/dL.
* Pregnancy or breastfeeding.
* History of hypersensitivity to hydrochlorothiazide or furosemide.
* Patients admitted from the Intensive Care Unit.
* Patients with recent cardiac surgery (within the last year) or heart transplant recipients.
* Need for inotropic support to maintain adequate cardiac and/or renal output.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2025-03-10 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Significant reduction in congestion (ADVOR scale) | After the first 72 hours of endovenous loop diuretic treatment
  To evaluate the significant reduction in congestion (ADVOR Scale) after the first 72 hours of intravenous diuretic treatment in the hospital ward, comparing the standard treatment group with the intervention group (intra-abdominal pressure and ultrasound).
  ADVOR Scale:
  Oedema: No oedema (0 points), Trace oedema (1 point), Clear pitting oedema (2 points), Visual deformation above ankle (3 points), Visual deformation above knee (4 points).
  Pleural effusion: No pleural effusion (0 points), Minor (2 points), Major (3 points)
  Ascites: No ascites (0 points), Minor ascites (2 points), Significant ascites (3 points)
  TOTAL SCORE: Oedema score + Pleural effusion + Ascitis. Minimum 0 points; Maximum 10 points

SECONDARY OUTCOMES:
Significant pulmonary congestion reduction through lung ultrasound assessment (b-lines) | From time to randomization until the first 72 hours of endovenous loop diuretics treatment at the Internal Medicine ward
  To evaluate the complete resolution of pulmonary congestion as assessed by ultrasound (B-lines) after the first 72 hours of intravenous diuretic treatment in the hospital ward, comparing the standard of care treatment group with the interventional group (intra-abdominal pressure and ultrasound).
  The degree of pulmonary tissue congestion will be quantified using clinical ultrasound. Eight quadrants (four left and four right) will be examined. A quadrant will be considered positive for pulmonary tissue congestion if three or more B-lines are detected. Minimum: 0 quadrants; Maximum 8 quadrants
Significant intravascular congestion reduction through venous excess ultrasound score (VEXUS score) | After the first 72 hours of endovenous loop diuretic treatment
  To evaluate the significant reduction in intravascular congestion (inferior vena cava diameter and venous excess ultrasound protocol) after the first 72 hours of intravenous diuretic treatment in the hospital ward, comparing the standard of care treatment group with the interventional group (intra-abdominal pressure and ultrasound).
  VEXUS score
  * Grade 0: No congestion; inferior vena cava vein (IVC) diameter < 2 cms
  * Grade 1: Mild congestion, IVC 2> cms + any combination of normal or mildly abnormal waveforms of doppler veins explored.
  * Grade 2: Moderate congestion, IVC > 2 cms + at least one severely abnormal pattern of doppler veins explored.
  * Grade 3: Severe congestion, IVC > 2cms + two or more severely abnormal waveforms of doppler veins explored.
  Minimum 0 points; Maximum 3 points
Total diuresis response | After the first 72 hours of endovenous loop diuretic treatment
  To evaluate the diuretic response (total urine volume/total dose of furosemide administered) after the first 72 hours of intravenous diuretic treatment in the hospital ward, comparing the standard treatment group with the intervention group (intra-abdominal pressure and ultrasound).
Total dose of diuretic treatment | After the first 72 hours of endovenous loop diuretic treatment
  To compare the days and doses of intravenous loop diuretics and hydrochlorothiazide used during the first 72 hours of hospitalization between the standard treatment group and the intervention group.
Number of patients treated for worsening heart failure | From date of discharge until 30-days post-hospitalization visit. From date of discharge until 90-days post-hospitalization visit. (cut-off period 1-year)
  Differences in heart failure worsening (defined as the need for intravenous loop diuretic treatment after hospital discharge, whether in a day hospital, emergency department, or due to new hospital admissions at 30 and 90 days) between the two groups.
Total number of patients with cardiovascular death | From date of discharge until the date of cardiovascular death (cut-off period 1 year)
  Differences in cardiovascular death incidence
guided directed medical therapy (GDMT) | From date of admission up to discharge, from date of discharge up to 30 days after and from date of discharge up to 90 days (cut-off period 1-year)
  Prevalence of GDMT prescribed at discharge according to left ventricular ejection fraction and actual heart failure guidelines
length of stay | From date of randomization until date of discharge (cut-off period 4 weeks)
  Differences in length of stay between both arms

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clínico Universitario Lozano Blesa, Zaragoza, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Website of the Spanish Medicines Agency where the clinical trial is registered in clinical trial information system (CTIS) — https://reec.aemps.es/reec/public/detail.html